CLINICAL TRIAL: NCT04616040
Title: A Non-interventional Registration Study Evaluating the Usage of Camrelizumab in the Treatment of Unresectable Locally Advanced/Recurrent or Metastatic Chinese Patients With Esophageal Cancer
Brief Title: A Real-world Study Evaluating the Usage of Camrelizumab in Chinese Patients With Advanced Esophageal Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Professor, Peking University
Other Study IDs: LION-EC
Record Dates: First submitted 2020-10-10; First posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — camrelizumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- unresectable locally advanced/recurrent or metastatic esophageal cancer
  Interventions: Drug: Camrelizumab

INTERVENTIONS:
Drug: Camrelizumab — The recommended formulation of Camrelizumab is 200 mg every time, or 3 mg/Kg according to body weight, intravenously infused.

SUMMARY:
The trial is a multi-center, open, observational registration study, which aims to evaluate the safety and efficacy of Camrelizumab (anti-PD-1 antibody) in the treatment of Chinese patients with advanced esophageal cancer in the real world.

ELIGIBILITY:
Inclusion Criteria:

1. Sign informed consent and voluntarily participate in this study.
2. Unresectable locally advanced/recurring or distant metastatic esophageal cancer patients confirmed by histology or cytology (AJCC 8th edition);

   * Unresectable locally advanced patients who are unable or unable to receive radical treatment (including radical radio chemotherapy or radical radiotherapy, etc.) may be considered for inclusion;
   * Patients who progress or relapse after neoadjuvant or adjuvant therapy may also be considered for inclusion;
3. Age ≥ 18 years old;
4. The investigator determines that the patient can receive Camrelizumab as a single agent or combination therapy.

Exclusion Criteria:

1. Evidence suggests that the patient is pregnant or breastfeeding;
2. Other drug blinded clinical trials are currently underway;
3. Other situations that are not suitable for inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: unresectable locally advanced/recurrent or metastatic esophageal cancer
Sampling Method: Probability Sample
Enrollment: 1030 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events of Camrelizumab | an expected average of 24 months
  especially Occurrence of ≥Grade 3 immune-related AEs

SECONDARY OUTCOMES:
Adverse events of Camrelizumab | an expected average of 24 months
  including other occasional or rare AEs
Overall Survival | an expected average of 24 months
  Duration from the date of initial treatment to the date of death due to any cause
Progression-free Survival (PFS) | an expected average of 24 months
  A duration from the date of initial treatment to radiographic disease progression or death of any cause
Objective Response Rate (ORR) | an expected average of 24 months
  Proportion of objective complete response and partial response patients

OTHER OUTCOMES:
Correlations between biomarkers and clinical activity | an expected average of 24 months
  tumor biopsies are collected before start of treatment, for assessing the relationship between different biomarkers (e.g. PD-L1 expression) with different camrelizumab-based regimens

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China